CLINICAL TRIAL: NCT02940054
Title: Validation of the RED-FLAGS Index for Early Diagnosis of Crohn's Disease: Prospective Observational Study
Brief Title: RED-FLAGS Index Validation in Crohn's Disease Patients
Acronym: RED-FLAGS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Takeda (Industry); IG-IBD talian Group for Inflammatory Bowel Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1414
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease
Keywords: Early diagnosis
MeSH Terms: conditions — Crohn Disease; Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patents with suspected Crohn's disease: Adult patients showing at least one of the following symptoms, from at least 4 weeks:
  * diarrhea
  * nocturnal diarrhea
  * body weight loss (>5%)
  * abdominal pain
  * perianal lesions.
  Interventions: Other: Red-flags questionnaire

INTERVENTIONS:
Other: Red-flags questionnaire — A questionnaire composed by 8 items will be administered by GPs to those patients and they will be referred to a gastroenterologist with expertise in CD. All those patients will be evaluated, as per usual practice, to confirm or exclude Crohn's disease.

SUMMARY:
Observational prospective study to validate a new index for early diagnosis of Crohn's disease (CD)

DETAILED DESCRIPTION:
The study will be conducted in Italian referral centers for Crohn's disease and will involve general practitioners (GPs) for RED-Flags Index validation.

The project is divided into two phases.

1. retrospective phase (4 weeks). All the general practitioners participating to the study will extrapolate from their patient's database, the total number of patients with a Crohn's disease diagnosis performed in the past. The date of diagnosis will be indicated. No other information will be provided. These data will be then analyzed to obtain, for each GP, the total number of CD diagnosed in each semester.
2. retrospective phase (6 months). GPs will administer the RED-Flags questionnaire to all patients that meet inclusion and exclusion criteria, after informed consent signature. All these patients will be then referred to the nearest referral center, to be evaluated by a gastroenterologist specialized in CD, to confirm or exclude a CD.

ELIGIBILITY:
Inclusion Criteria:

1. at least one of the following symptoms, for at least 4 weeks (either continuous or intermittent)

   1. diarrhea (>3 bowel movements per day)
   2. nocturnal diarrhea
   3. weight loss (≥5% of usual body weight)
   4. abdominal pain (chronic or intermittent)
   5. perianal lesions or fistulae or perianal abscess (hemorrhoidal diseases excluded)
2. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements. The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. known diagnosis of Crohn's disease, ulcerative colitis, chronic diverticulosis or any other gastrointestinal disease
2. any clinical condition that, in the opinion of the investigator, can alter stud results
3. inability to understanding and complying with protocol requirements
4. informed consent not signed and dated by the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 subjects, aged 18-65, requiring general practitioner's advise for gastrointestinal symptoms compatible with Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Sensibility of the Red Flags Index | at enrollment
  Sensibility, specificity, accuracy, positive and negative likelihood ratio measurement

SECONDARY OUTCOMES:
Percentage of early diagnosed | 6 months of prospective period
  Percentage of early diagnosed of Crohn's Disease in the 6 months of prospective use of the tool
Cut-off for Crohn's disease diagnosis | at enrollment
  Identification of the cut-off associated with an early diagnosis of Crohn's disease

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Gavazzeni, Bergamo, BG, Italy

REFERENCES:
- [Background] Danese S, Fiorino G, Mary JY, Lakatos PL, D'Haens G, Moja L, D'Hoore A, Panes J, Reinisch W, Sandborn WJ, Travis SP, Vermeire S, Peyrin-Biroulet L, Colombel JF. Development of Red Flags Index for Early Referral of Adults with Symptoms and Signs Suggestive of Crohn's Disease: An IOIBD Initiative. J Crohns Colitis. 2015 Aug;9(8):601-6. doi: 10.1093/ecco-jcc/jjv067. Epub 2015 Apr 23. PMID 25908718